CLINICAL TRIAL: NCT06158243
Title: Description of the Brachial Plexus Block at the Humeral Head in Children: a Sono-anatomical Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Raoul Ngatcha, MD, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: B062023230501
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia, Local; Brachial Plexus; Pressure
Keywords: Brachial plexus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 0-2: children aged 0 to 2 years
  Interventions: Other: Sono-anatomical Study
- 2-4: children aged 2 to 4 years
- 4-6: children aged 4 to 6 years
- 6-8: children aged 6 to 8 years
  Interventions: Other: Sono-anatomical Study
- 8-10: children aged 8 to 10 years

INTERVENTIONS:
Other: Sono-anatomical Study — The arm is abducted (90°), externally rotated, with the forearm flexed over the arm (90°). A linear ultrasound probe (8-15 MHz) is placed in front of the humeral head, in a sagittal plane. Location begins at axillary level, vessels, nerves and humerus are identified, and the probe is moved medially to reach and identify the humeral head.
  Groups: 0-2; 6-8

SUMMARY:
the investigators are interested in assessing the feasibility and value of brachial plexus block at the level of the humeral head in children. As a first step, the investigators propose to carry out a sono-anatomical study to describe the plexus at this level, the distribution of nerves in relation to the axillary artery, and the description of bone and muscle structures.

DETAILED DESCRIPTION:
Brachial plexus blocks below the clavicle provide anesthesia and analgesia of the upper limb for elbow, forearm and hand surgery. Among the techniques described, axillary and costo-clavicular blocks are most frequently used.

In the axillary approach to the brachial plexus, the ulnar, median and radial nerves are in the direct vicinity of the axillary artery. However, there is considerable variability in the location of these nerves . What's more, the musculocutaneous nerve is most often distant from the other nerves of the plexus. These disadvantages are not encountered with the costo-clavicular technique, in which the nerves are brought together in the same diffusion space. On the other hand, this method does run the risk of pneumothorax and anesthesia of the phrenic nerve.

In this context, the investigators have described the brachial plexus block at the level of the humeral head in adults, which enables practicians to work on nerves gathered around the axillary artery without any risk of phrenic or pulmonary damage4.

In children, Small et al described a supra-clavicular approach, but Clayton et al, noting the high risk of pneumothorax, strongly advocated the axillary approach.

ELIGIBILITY:
Inclusion Criteria:

* patient ASA 1-2
* aged 0 to 10 years
* scheduled surgery
* parental consent obtained

Exclusion Criteria:

* Parental refusal to participate
* suspicion of local skin infection
* inability to place the limb in the position required for sonographic examination
* Upper limb malformation
* ASA III, IV
* Major surgery (cardiac, neurosurgery...)
* emergencies

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be carried out in 100 children aged 0-10, divided into 5 groups of 20: 0-2 years, 2-4 years, 4-6 years, 6-8 years and 8-10 years. After obtaining informed consent from parents, patients will be included in the study according to inclusion and exclusion criteria. Sonographic observations and measurements will be performed during narcosis, if possible, without delaying or interfering with surgery. No puncture will be performed.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
description of the position of the nerves around the axillary artery | through study completion, around 5 months
  Hourly distribution of nerve structures around the axillary artery , expressed in degrees and measured with a protractor

SECONDARY OUTCOMES:
distance between anatomical structures | through study completion, around 5 months
  depth of diffusion spaces Skin-cartilage distance Cartilage thickness Skin-nerve distance Skin-to-vessel distance size of nerves all these measurements in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GUNTZ, Study Director — Anesthesiologist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nalini KB, Bevinaguddaiah Y, Thiyagarajan B, Shivasankar A, Pujari VS. Ultrasound-guided costoclavicular vs. axillary brachial plexus block: A randomized clinical study. J Anaesthesiol Clin Pharmacol. 2021 Oct-Dec;37(4):655-660. doi: 10.4103/joacp.JOACP_43_20. Epub 2021 Nov 2. PMID 35340944
- [Background] Christophe JL, Berthier F, Boillot A, Tatu L, Viennet A, Boichut N, Samain E. Assessment of topographic brachial plexus nerves variations at the axilla using ultrasonography. Br J Anaesth. 2009 Oct;103(4):606-12. doi: 10.1093/bja/aep207. Epub 2009 Aug 21. PMID 19700445
- [Background] SMALL GA. Brachial plexus block anesthesia in children. J Am Med Assoc. 1951 Dec 22;147(17):1648-51. doi: 10.1001/jama.1951.03670340038009. No abstract available. PMID 14880419
- [Background] Li JW, Songthamwat B, Samy W, Sala-Blanch X, Karmakar MK. Ultrasound-Guided Costoclavicular Brachial Plexus Block: Sonoanatomy, Technique, and Block Dynamics. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):233-240. doi: 10.1097/AAP.0000000000000566. PMID 28157792
- See also: this work is the first we have done in adults " brachial intermediate nerve block" — https://rapm.bmj.com/content/47/Suppl_1/A126.1